CLINICAL TRIAL: NCT01631604
Title: Quantification of Gait Parameters and Muscle Activation Patterns Following a Fall
Brief Title: Gait Characteristics Following a Fall
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Model: Factorial | Purpose: Treatment
Other Study IDs: Fall-HMO-CTIL
Record Dates: First submitted 2012-06-28; First posted 2012-06-29 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2012-06

CONDITIONS: Motor Impairments; Orthopaedic Injuries; Neurological Conditions
Keywords: risk of falling; gait patterns; muscle activity; fall prevention; motor impairment
MeSH Terms: interventions — Equipment and Supplies; Botulinum Toxins; Bupivacaine; Meniscectomy; Anterior Cruciate Ligament Reconstruction; Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip; Physical Therapy Modalities

INTERVENTIONS:
Device: Walking aids and devices — Walking aids, e.g. braces, canes,orthoses, prosthetics, etc.
Drug: Muscle/nerve injection — Injection to muscle or nerve
  Other Names: Botulinum toxin; Marcaine
Procedure: Corrective surgery — correction of spinal and bony deformities, muscle transfer, tendon elongation etc.
  Other Names: Knee arthroscopy, meniscectomy and chondroplasty; Anterior cruciate ligament reconstruction; Knee replacement; Repair of femoral neck fracture; Repair of trochanteric fracture; Debridement of skin/muscle/bone/fracture; Knee arthroscopy repair of both menisci; Hip replacement; Repair of ankle fracture (bimalleolar type); Lumbar spinal fusion; Low back intervertebral disc surgery; Repair of femoral shaft fracture
Other: Physical therapy treatment

SUMMARY:
The purpose of this study is to quantify the safety degree of the patient's gait, to detect the reason for the fall and quantify the biomechanical parameters related to fall. This study also aims to evaluate the effect of different rehabilitation treatments and their effect on the risk of falling.

DETAILED DESCRIPTION:
In this study, patients suffering from motor disabilities as a result of orthopedic or neurologic impairments will be tested at the gait and motion laboratory. Each patient will be secured with a ceiling-mounted safety harness and will walk on the path wearing passive light-reflecting markers and surface electrodes. High-speed cameras will record the subject's movements and the markers will be tracked to produce data of joint angles, velocities and accelerations. Dynamic EMG will be recorded from various muscles.

During the examination, the gait of the subjects will be disturb by either (i) a visual or sound signal that requires the subject to stop immediately, or (ii) walking different terrains, or (iii) tying a string to the foot and pulling it shortly to induce a trip.

ELIGIBILITY:
Inclusion Criteria:

* Individuals suffering from gait impairment following injury to the central or peripheral nervous system, as well as following orthopedic injuries. The subjects will be able to understand and independently sign a consent form.

Exclusion Criteria:

* Subjects who are unable to understand and independently sign a consent form
* Subjects who are wheelchair bound.
* Pregnant women.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Gait kinematics
  Joint angles, velocities and accelerations

SECONDARY OUTCOMES:
Muscle activation patterns
  Dynamic EMG of various muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel